CLINICAL TRIAL: NCT03609099
Title: Adequate Duration of Antibiotic Treatment in Community-acquired Pneumonia With High Risk Class and Adequate Initial Clinical Response
Acronym: 2017-001406-15
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: David Garcia Cinca (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other); Miquel Ferrer - Investigator Coordinator (Unknown)
Responsible Party: Sponsor-Investigator, David Garcia Cinca, Study Applicant, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAC-ATB
Record Dates: First submitted 2018-07-23; First posted 2018-08-01 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moxifloxacin (Active Comparator): Active treatment to patients treated during the 5 previous days.
  Interventions: Drug: Moxifloxacin
- Placebo (Experimental): Placebo treatment to patients treated during the 5 previous days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Moxifloxacin — 400 mg / day once a day oral treatment during 3 days.
  Other Names: Active treatment
  Arms: Moxifloxacin
Drug: Placebo — once a day oral treatment during 3 days.
  Arms: Placebo

SUMMARY:
Non-inferiority, multicenter, prospective double-blind, randomized clinical trial of two parallel groups. The randomization between the 2 study groups will be carried out according to a scheme generated by a computer program, in blocks of 6 and stratified by centers. The antibiotic treatment will be evaluated during 5 days compared to the usual antibiotic treatment for more than 7 days in patients with community-acquired pneumonia with a Pneumonia Severity Index IV-V severity score who present an adequate response in the first 4 days of hospital antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes older than 18 years
* Hospitalized patients diagnosed with CAP: appearance of a new radiological infiltrate plus the presence of at least two of the following signs or symptoms: fever (> 38 ° C), cough, expectoration, chest pain, dyspnea or tachypnea, and signs of occupation of the alveolar space.
* That they present a PSI score class IV or V.
* Patients who have received adequate antibiotic treatment according to clinical guidelines (SEPAR, ATS) ((1,8,19)) from the first hour of admission to the emergency room.
* Patients who reach clinical stability: temperature ≤37.2 ºC, heart rate ≤100 beats / min, respiratory rate ≤24 breaths / min, systolic blood pressure> 90 mmHg; oxygen saturation> 90%; or oxygen blood pressure> 60 mmHg (15) before the fourth day.
* Signature of informed consent.

Exclusion Criteria:

* Immunosuppression: Co infection with HIV and presence of AIDS, treatment with neutropenic effect or have received immunosuppressive treatment for any reason. Patients that are in chronic use of corticosteroids as prednisone or its equivalent with > 10 mg / day for 14 days.
* Patients hospitalized in the previous 14 days.
* Patients with pleural effusion
* Suspected multiresistant germs of any cause.
* Hypersensitivity or alterations in the tendons associated with the fuoroquinolones.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
Rate of treatment failure | during the 30 days after the day of hospital admission
  Treatment failure is defined as the appearance of any of the following manifestations: death from any cause, hospital readmission for any cause or restart of antibiotic treatment for any reason.

SECONDARY OUTCOMES:
Length of hospital stay | up to 2 years
Antibiotic-free days | Up to 28 days
  Antibiotic-free days are defined as the number of days alive and free of antibiotics
Proportion of adverse events | Up to 28 days
Proportion of serious adverse events | Up to 28 days

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Galdakao-Usansolo, Galdakao, Bizkaia
  - Hospital Universitario La Fe, Valencia, Valencia
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Virgen de Valme, Seville